CLINICAL TRIAL: NCT00925470
Title: Evaluation of Target Organs Impairment on Patients Suffering From High Blood Pressure Without Known Cardio Vascular or Renal Disease, Stratified on Blood Pressure Control.
Brief Title: Evaluation of Target Organs Impairment on Patients Suffering From High Blood Pressure
Acronym: PREVENTA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CFR-DUM-2009/1
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2009-12-18 (Estimated); Status verified 2009-12

CONDITIONS: Blood Pressure
Keywords: Target organs impairment; High blood pressure; Evaluation of target organs impairment on patients suffering from high blood pressure without known cardiovascular or renal disease
MeSH Terms: conditions — Hypertension; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Evaluation of target organs impairment on patients suffering from high blood pressure without known cardio vascular or renal disease, stratified on blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Adults with hypertension (treated or not), without known cardiovascular or renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First 2 consecutive adults with hypertension, without known cardio vascular or renal disease,seen by Cardiologists
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2009-06; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the frequency of evaluation of target organs preclinical impairment on patients without known cardiovascular or renal disease, taking into consideration the blood pressure level (controlled HBP or not) | Once

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne, Medical Director, Study Director — AstraZeneca
Locations (369):
- France (369):
  - Research Site, Abbeville
  - Research Site, Aire-sur-l'Adour
  - Research Site, Aix-en-Provence
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Ambérieu-en-Bugey
  - Research Site, Ambilly
  - Research Site, Amiens
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Angers
  - Research Site, Angoulême
  - Research Site, Annecy
  - Research Site, Annemasse
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Apt
  - Research Site, Arbois
  - Research Site, Arles
  - Research Site, Armentières
  - Research Site, Asnières-sur-Seine
  - Research Site, Aubenas
  - Research Site, Aubervilliers
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Aulnay-sous-Bois
  - Research Site, Bagnères-de-Bigorre
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baie Mahault
  - Research Site, Bailleul
  - Research Site, Basse Terre
  - Research Site, Bastia
  - Research Site, Bayeux
  - Research Site, Beauchamp
  - Research Site, Beaumont
  - Research Site, Beaumont-de-Lomagne
  - Research Site, Beaumont-sur-Oise
  - Research Site, Beausoleil
  - Research Site, Beauvais
  - Research Site, Belfort
  - Research Site, Bellegarde-sur-Valserine
  - Research Site, Belley
  - Research Site, Bergerac
  - Research Site, Besançon
  - Research Site, Béthune
  - Research Site, Béziers
  - Research Site, Biscarrosse
  - Research Site, Blaye
  - Research Site, Bobigny
  - Research Site, Bois-Colombes
  - Research Site, Bois-Guillaume
  - Research Site, Bordeaux
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourges
  - Research Site, Bourgoin
  - Research Site, Brest
  - Research Site, Brive-la-Gaillarde
  - Research Site, Bron
  - Research Site, Brunoy
  - Research Site, Bry-sur-Marne
  - Research Site, Bussy-Saint-Georges
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cahors
  - Research Site, Caluire-et-Cuire
  - Research Site, Cambo-les-Bains
  - Research Site, Carcassonne
  - Research Site, Carpentras
  - Research Site, Carquefou
  - Research Site, Castanet-Tolosan
  - Research Site, Castelnau-le-Lez
  - Research Site, Castelnaudary
  - Research Site, Castelsarrasin
  - Research Site, Castres
  - Research Site, Cenon
  - Research Site, Cergy
  - Research Site, Chambéry
  - Research Site, Chamonix
  - Research Site, Champigny-sur-Marne
  - Research Site, Charleville-Mézières
  - Research Site, Chartres
  - Research Site, Chatou
  - Research Site, Châlons-en-Champagne
  - Research Site, Château-d'Olonne
  - Research Site, Château-Thierry
  - Research Site, Châteaubernard
  - Research Site, Châteauroux
  - Research Site, Châtillon-sur-Seine
  - Research Site, Chelles
  - Research Site, Cherbourg Octeville
  - Research Site, Clermont-Ferrand
  - Research Site, Compiègne
  - Research Site, Condé-sur-l'Escaut
  - Research Site, Conflans Ste Honorine
  - Research Site, Coubron
  - Research Site, Courbevoie
  - Research Site, Coutances
  - Research Site, Creil
  - Research Site, Croix
  - Research Site, Dax
  - Research Site, Deauville
  - Research Site, Denain
  - Research Site, Décines-Charpieu
  - Research Site, Dieppe
  - Research Site, Dijon
  - Research Site, Dinard
  - Research Site, Divion
  - Research Site, Dole
  - Research Site, Domont
  - Research Site, Douai
  - Research Site, Draguignan
  - Research Site, Dunkirk
  - Research Site, Elbeuf
  - Research Site, Enghien-les-Bains
  - Research Site, Esbly
  - Research Site, Échirolles
  - Research Site, Épernay
  - Research Site, Épinal
  - Research Site, Étampes
  - Research Site, Évecquemont
  - Research Site, Évreux
  - Research Site, Faches-Thumesnil
  - Research Site, Firminy
  - Research Site, Floirac
  - Research Site, Fontaine
  - Research Site, Fontainebleau
  - Research Site, Fontenay-sous-Bois
  - Research Site, Fort de France
  - Research Site, Fougères
  - Research Site, Fourmies
  - Research Site, Frontignan
  - Research Site, Gagny
  - Research Site, Gap
  - Research Site, Garches
  - Research Site, Gasville-Oisème
  - Research Site, Genas
  - Research Site, Gennevilliers
  - Research Site, Gien
  - Research Site, Givet
  - Research Site, Givors
  - Research Site, Gleizé
  - Research Site, Gourdon
  - Research Site, Gray
  - Research Site, Grenoble
  - Research Site, Guebwiller
  - Research Site, Guéret
  - Research Site, Guilherand-Granges
  - Research Site, Hagondange
  - Research Site, Haguenau
  - Research Site, Hesdin
  - Research Site, Héricourt
  - Research Site, Hérouville-Saint-Clair
  - Research Site, Hyères
  - Research Site, Issy-les-Moulineaux
  - Research Site, Ivry-sur-Seine
  - Research Site, Jonzac
  - Research Site, Juan-les-Pins
  - Research Site, Juvisy-sur-Orge
  - Research Site, L'Isle-sur-la-Sorgue
  - Research Site, La Garenne-Colombes
  - Research Site, La Madeleine
  - Research Site, La Seyne-sur-Mer
  - Research Site, Lamotte-Beuvron
  - Research Site, Lanester
  - Research Site, Langon
  - Research Site, Lannemezan
  - Research Site, Lannion
  - Research Site, LArbresle
  - Research Site, Le Chesnay
  - Research Site, Le Havre
  - Research Site, Le Mans
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Pontet
  - Research Site, Le Port
  - Research Site, Le Port-Marly
  - Research Site, Le Relecq-Kerhuon
  - Research Site, Le Tampon
  - Research Site, Lens
  - Research Site, Les Ulis
  - Research Site, Lesparre-Médoc
  - Research Site, Levallois-Perret
  - Research Site, Liévin
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Limoux
  - Research Site, Lisieux
  - Research Site, Livry-Gargan
  - Research Site, Longjumeau
  - Research Site, Loos
  - Research Site, Lorient
  - Research Site, Lunel
  - Research Site, Lyon
  - Research Site, Mainvilliers
  - Research Site, Maisons-Alfort
  - Research Site, Marck En Baroeul
  - Research Site, Marmande
  - Research Site, Maromme
  - Research Site, Marseille
  - Research Site, Marvejols
  - Research Site, Massy
  - Research Site, Maubeuge
  - Research Site, Melun
  - Research Site, Mende
  - Research Site, Mennecy
  - Research Site, Metz
  - Research Site, Mérignac
  - Research Site, Millau
  - Research Site, Mont-de-Marsan
  - Research Site, Montargis
  - Research Site, Montauban
  - Research Site, Montbéliard
  - Research Site, Montbrison
  - Research Site, Montmorillon
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montrouge
  - Research Site, Morlaix
  - Research Site, Nancy
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Neufchâteau
  - Research Site, Nevers
  - Research Site, Nice
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Noisy-le-Sec
  - Research Site, Noyon
  - Research Site, Oignies
  - Research Site, Olivet
  - Research Site, Ollioules
  - Research Site, Orléans
  - Research Site, Orly
  - Research Site, Orthez
  - Research Site, Pamiers
  - Research Site, Pantin
  - Research Site, Paray-le-Monial
  - Research Site, Paris
  - Research Site, Pau
  - Research Site, Perpignan
  - Research Site, Péronne
  - Research Site, Pierrelatte
  - Research Site, Pithiviers
  - Research Site, Plaisance-du-Touch
  - Research Site, Ploërmel
  - Research Site, Pointe à Pitre
  - Research Site, Poitiers
  - Research Site, Pompey
  - Research Site, Pont-à-Mousson
  - Research Site, Pont-d'Héry
  - Research Site, Pontarlier
  - Research Site, Pontault-Combault
  - Research Site, Pontcharra
  - Research Site, Pontoise
  - Research Site, Prades
  - Research Site, Prévessin-Moëns
  - Research Site, Puilboreau
  - Research Site, Quimperlé
  - Research Site, Quincy-sous-Sénart
  - Research Site, Rambouillet
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Revel
  - Research Site, Rillieux-la-Pape
  - Research Site, Rixheim
  - Research Site, Rodez
  - Research Site, Romans-sur-Isère
  - Research Site, Romorantin-Lanthenay
  - Research Site, Rosny-sous-Bois
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Royan
  - Research Site, Royat
  - Research Site, Sablé-sur-Sarthe
  - Research Site, Saint-Amand-Montrond
  - Research Site, Saint-André-les-Vergers
  - Research Site, Saint-Avold
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Chamond
  - Research Site, Saint-Dié
  - Research Site, Saint-Etienne
  - Research Site, Saint-Flour
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Saint-Herblain
  - Research Site, Saint-Ismier
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Leu
  - Research Site, Saint-Louis
  - Research Site, Saint-Martin-Boulogne
  - Research Site, Saint-Martin-d'Aubigny
  - Research Site, Saint-Martin-d'Hères
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pol-de-Léon
  - Research Site, Saint-Pol-sur-Mer
  - Research Site, Saint-Quentin
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Renan
  - Research Site, Saint-Yrieix-la-Perche
  - Research Site, Saintes
  - Research Site, Salon-de-Provence
  - Research Site, Sanary-sur-Mer
  - Research Site, Sarcelles
  - Research Site, Sarreguemines
  - Research Site, Saumur
  - Research Site, Savigny-sur-Orge
  - Research Site, Schiltigheim
  - Research Site, Sevran
  - Research Site, Sète
  - Research Site, Sélestat
  - Research Site, Six-Fours-les-Plages
  - Research Site, Somain
  - Research Site, Sorgues
  - Research Site, Stains
  - Research Site, Ste Clotilde Cedex
  - Research Site, Ste Foy La Grande
  - Research Site, Strasbourg
  - Research Site, Suresnes
  - Research Site, Talence
  - Research Site, Tarbes
  - Research Site, Taverny
  - Research Site, Tergnier
  - Research Site, Ternay
  - Research Site, Thann
  - Research Site, Thionville
  - Research Site, Thouars
  - Research Site, Tonneins
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tournefeuille
  - Research Site, Tournon-sur-Rhône
  - Research Site, Tours
  - Research Site, Tracy-le-Mont
  - Research Site, Trappes
  - Research Site, Triel-sur-Seine
  - Research Site, Troyes
  - Research Site, Ussel
  - Research Site, Valence
  - Research Site, Valenciennes
  - Research Site, Valognes
  - Research Site, Valréas
  - Research Site, Vanves
  - Research Site, Vence
  - Research Site, Vendôme
  - Research Site, Vernon
  - Research Site, Verrières-le-Buisson
  - Research Site, Versailles
  - Research Site, Vénissieux
  - Research Site, Vichy
  - Research Site, Vierzon
  - Research Site, Vigneux-sur-Seine
  - Research Site, Ville-d'Avray
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villejuif
  - Research Site, Villeneuve Saint Georges Cede
  - Research Site, Villeneuve-sur-Lot
  - Research Site, Villepinte
  - Research Site, Villeurbanne
  - Research Site, Villiers-sur-Orge
  - Research Site, Vincennes
  - Research Site, Vitré
  - Research Site, Wattignies
  - Research Site, Yvetot